CLINICAL TRIAL: NCT03306836
Title: Multi-center，Single Blind，Prospective Randomized Controlled Trial of Exploration of Anticoagulation Program in Cerebral Aneurysm and Arteriovenous Malformations With Hybrid Operation
Brief Title: Exploration of Anticoagulation Program in Cerebral Aneurysm and Arteriovenous Malformations With Hybrid Operation 2
Acronym: EAPCAAMHO2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Tang-Du Hospital (Other); Kunming Medical University (Other); First Affiliated Hospital of Fujian Medical University (Other); Nanjing PLA General Hospital (Other); Fujian Medical University Union Hospital (Other)
Responsible Party: Principal Investigator, Dr. Yong Cao, principal, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016YFC1301800-2
Record Dates: First submitted 2017-05-31; First posted 2017-10-11 (Actual); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Cerebral Aneurysm; Arteriovenous Malformations
Keywords: Hybrid operation; Cerebral Aneurysm; Arteriovenous Malformations; Anticoagulation
MeSH Terms: conditions — Intracranial Aneurysm; Arteriovenous Malformations | interventions — Heparin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard dose group of Heparin Sodium (Experimental): First infused with 5000 IU of Heparin Sodium, then continuous infusion at a rate of 18 IU / kg.h during the hybrid operation.
  Interventions: Drug: Heparin Sodium
- Low dose group of Heparin Sodium (Active Comparator): infusion Heparin Sodium at a rate of 18 IU / kg.h during the hybrid operation.
  Interventions: Drug: Heparin Sodium

INTERVENTIONS:
Drug: Heparin Sodium — Infused with 5000 IU of Heparin Sodium
  Arms: Standard dose group of Heparin Sodium
Drug: Heparin Sodium — Infusion Heparin Sodium at a rate of 18 IU / kg.h

SUMMARY:
In the stage of randomized controlled study, our purpose is to obtain the Intraoperative anticoagulation program supported by evidence-based medicine.

DETAILED DESCRIPTION:
This study is divided into anticoagulation program in cerebral aneurysm with hybrid operation and anticoagulation program in cerebral arteriovenous malformations with hybrid operation two parts, and each part divide into two stage, on the stage of registration study. This study is a multi-center, single-blind, prospective cohort study. Record the patient's intraoperative activated coagulation time Changes in detail, to observe the effect of activated coagulation time maintenance level on hemorrhage event rate of Intraoperative and postoperative 48 hours, purpose to find out the safety range of activated coagulation time level in cerebral aneurysm and arteriovenous malformations with hybrid operation. On the stage of randomized controlled study. This study is a multicenter, single-blind, prospective, randomized controlled study. Patients is divided into intraoperative standard dose group of Heparin Sodium and low dose group of Heparin Sodium randomly. To observe the effect of different anticoagulation regimens on activated coagulation time safety coverage rate during surgery, and finally develop a scientific and effective intraoperative anticoagulant therapy program.

ELIGIBILITY:
Inclusion Criteria:

1.All patients undergoing hybird surgery.

Exclusion Criteria:

1. Poor general condition , severe primary disease, surgical contraindications
2. Patient or family refused surgery
3. Fusiform aneurysm,Traumatic aneurysm,Infectious aneurysms
4. Combined with other hemorrhagic cerebrovascular disease
5. Combined with malignant brain tumor
6. Perinatal, Pregnancy
7. Patients unwilling to participate in the trial

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 408 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Changes in activated coagulation time safety coverage rate from the beginning of surgery to 48 hours after surgery | From the beginning of surgery to 48 hours after surgery
  Activated coagulation time average value falls in the safety coverage rate from the beginning of surgery to 48 hours after surgery.

SECONDARY OUTCOMES:
Changes in hemorrhage event rate from the beginning of surgery to 48 hours after surgery | From the beginning of surgery to 48 hours after surgery
  Hemorrhage event include intracranial hemorrhage caused by non-surgical reasons, as well as other organs or parts of the massive bleeding or small bleeding, Including subperitoneal hemorrhage, intraocular hemorrhage, gross hematuria, epistaxis time prolonged or repeated, gastrointestinal bleeding, hemoptysis, subconjunctival hemorrhage, hematoma greater than 5cm, bleeding difficult to control the and so on.
Changes in ischemia event rate from the beginning of surgery to 48 hours after surgery | From the beginning of surgery to 48 hours after surgery
  Ischemia event include Cerebral infarction and transient ischemic attack.
Intraoperative blood loss | From the beginning of surgery to 48 hours after surgery
  All the blood lost during the surgery should be collected and measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No